CLINICAL TRIAL: NCT05403320
Title: An Innovative Cuff Pressure Control and Evacuation of Subglottic Secretions To Prevent Pneumonia. A Multicenter Cluster-Randomized Trial
Brief Title: Cuff Pressure Control and Evacuation of Subglottic Secretions To Prevent Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4739
Record Dates: First submitted 2022-05-16; First posted 2022-06-03 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Multicenter cluster randomized controlled and open-label trial. Because intubation is an urgent intervention in critically ill patients patients with acute respiratory failure, individual randomization is considered too complex and we predetermined cluster of 9 consecutive patients, stratified by centers, with each cluster being assigned to one of the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AnapnoGuard group (Experimental): Patients intubated with AnapnoGuard endotracheal tube (polyvinylchloride tube with ellipsoidal shape, thin wall polyurethane cuff with dual suction lines and an extra venting line) which is connected to AnapnoGuard 100 System
  Interventions: Device: Continuous cuff pressure regulation; Device: Automatic subglottic secretion drainage; Diagnostic Test: Tracheobronchial colonization assessment; Diagnostic Test: Microaspiration assessment; Diagnostic Test: VAP assessment
- Control group (Active Comparator): Patients intubated with TaperGuard Evac endotracheal tube (polyvinylchloride conic cuff with additional lumen for subglottic secretion suctioning)
  Interventions: Device: Intermittent cuff pressure regulation; Device: Manual subglottic secretion drainage; Diagnostic Test: Tracheobronchial colonization assessment; Diagnostic Test: Microaspiration assessment; Diagnostic Test: VAP assessment

INTERVENTIONS:
Device: Continuous cuff pressure regulation — Within 24 hours, AnapnoGuard tube will be connected to AnapnoGuard 100 control device. It includes an automatic high-sensitive subglottic capnograph which measures every few minutes the carbon dioxide level in the subglottic space. If the level of carbon dioxide is above the threshold (established by animal studies) the system will increase the cuff pressure by a formula, if the level is below the threshold, the system will decrease the cuff pressure by 1 mmHg. Variations of cuff pressure are allowed only between pressure limits set by the user (minimum and maximum)
  Arms: AnapnoGuard group
Device: Intermittent cuff pressure regulation — ET cuff pressure will be manually measured three times per day using a portable manometer, and kept constant within 20-30 cmH2O
  Arms: Control group
Device: Automatic subglottic secretion drainage — Within 24 hours, AnapnoGuard tube will be connected to AnapnoGuard 100 device control which provides continuous subglottic secretion drainage (two different suction lines) and venting/rinsing (a third dedicated line)
  Arms: AnapnoGuard group
Device: Manual subglottic secretion drainage — Subglottic secretions will be manually drained with a 10 mL syringe, using the only dedicated lumen
  Arms: Control group
Diagnostic Test: Tracheobronchial colonization assessment — Tracheal aspirate will be performed after intubation and after 72 hours for microbiological colture
Diagnostic Test: Microaspiration assessment — Tracheal aspirates will be performed 72 hours after intubation, and collected in a predefined study center to measure pepsin and salivary amylase
Diagnostic Test: VAP assessment — Patients will be follow to detect clinical, radiological or microbiological signs of VAP. If suspected, a tracheal aspirate or a bronchoalveolar lavage is performed to confirm the diagnosis

SUMMARY:
Multicenter, cluster randomized, controlled, open-label trial to assess if AnapnoGuard System can minimize tracheal microaspiration and the risk of ventilator-associated pneumonia when compared to standard treatment

DETAILED DESCRIPTION:
Maintaining the endotracheal tube (ETT) cuff appropriately inflated plays a crucial role in the management of intubated patients because overinflation may cause tracheal wall damage, ulcerations and stenosis, and underinflation may results in fluid leakage and ventilator-associated pneumonia (VAP).

During mechanical ventilation, secretions contaminated with oropharyngeal and gastric pathogens pool in the subglottic space (tracheal region between the ETT cuff and the vocal cords) and enter the lower airways via microaspiration.

Subglottic secretion drainage (SSD) reduces the incidence of VAP and can be performed intermittently or continuously, with varying efficacy and often causing secondary tracheal mucosa lesions.

AnapnoGuard (AG) ETT has three dedicated lines (two suction lines and one sensing/venting/rinsing line) and can be connected to the AG 100 System, a new device which provides high-sensitive capnography of subglottic space and consequent adjustment of cuff pressure, to avoid fluid leakage and overinflation. It also evacuates secretions from the subglottic space by simultaneously rinsing/venting this space using the ETT dedicated line.

The hypothesis is that AG System may reduce the incidence of microaspiration, bacterial tracheal colonization and consequently the risk of VAP when compared to standard treatment (ETT with manually performed secretion drainage and cuff pressure control).

ELIGIBILITY:
Inclusion Criteria:

* Primary intubation with the study ETT
* Expected duration of mechanical ventilation >48 hours
* Age older than 18 years

Exclusion Criteria:

* Invasive mechanical ventilation in the last 14 days,
* Contraindication for enteral feeding
* Clinical evidence of inhalation before intubation
* Pregnancy
* Enrolling in another study that may interfere with this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Bacterial tracheobronchial colonization (number of events) | 3 days
  The proportion of patients with bacterial tracheobronchial colonization (> 10^3 CFU/mL) on Day 3 after randomization, measured from tracheal aspirate

OTHER OUTCOMES:
Ventilator-associated pneumonia (number of events) | 28 days
  The proportion of patients who develop ventilator-associated pneumonia (presence of radiological and clinical signs consisting of a new and persistent infiltrate on the chest radiograph associated with two of the three following criteria: purulent tracheal aspirates, hyperthermia >38 °C or hypothermia <36 °C and peripheral leucocytosis >10,000/μ l or <1,500/μ. A microbiological confirmation is required using tracheal aspirate ≥ 10^5 CFU/ml or bronchoalveolar lavage ≥ 10^4 CFU/ml)
Microaspiration (number of events) | 2 days
  The prevalence of patients with gastric and oropharyngeal microaspiration or abundant microaspiration (Microaspiration is defined by the presence of alpha-amylase >1685 UI/L in tracheal aspirates. Abundant microaspiration is defined by pepsin level >200 ng/mL in >30 % of tracheal aspirates during the 48 h following inclusion.)
Ventilator-associated events (number of events) | 28 days
  The proportion of patients who develop ventilator-associated events, defined as a sustained increase in ventilator support (minimum PEP increase >2.5 cm H2 O, or minimum FiO2 increase >15 %) after >2 days of stable or decrease settings
Time to ventilator-associated pneumonia (days) | 28 days
  The time until the first diagnosis of ventilator-associated pneumonia is established
Antibiotic-free days (days) | 28 days
  The number of days in which the patient is not treated with any antibiotic drug
Ventilator-free days (days) | 28 days
  The number of days in which patients do not receive mechanical ventilation within 28 days from randomization
Length of intensive care unit stay (days) | 28 days
  The number of days in which the patient is admitted in intensive care unit or in hospital
Length of hospital stay (days) | 28 days
  The number of days in which the patient is admitted in hospital
In-intensive care unit mortality (number of events) | 28 days
  All-cause mortality, assessed at the discharge from the intensive care unit
In-hospital mortality (number of events) | 28 days
  All-cause mortality, assessed at the discharge from the hospital
28-day mortality (number of events) | 28 days
  All-cause 28-day mortality
60-day mortality (number of events) | 60 days
  All-cause 60-day mortality
90-day mortality (number of events) | 90 days
  All-cause 90-day mortality
Tracheobronchial colonization count (number of events) | 3 days
  The proportion of tracheal aspirates with colonization count >10^4, 10^5, 10^6, >= 10^7 CFU/mL
Post-extubation stridor (number of events) | 1 day
  The proportion of patients who experience stridor after extubation
Total subglottic secretion volume | 28 days
  The amount of secretions which has been drained from subglottic space during the enrolment
Daily subglottic secretion volume | 1 day
  Daily amount of secretions which has been drained from subglottic space
Out of range cuff pressure | 28 days
  The proportion of cuff pressure values whose are out of the safety limits

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro De Pascale, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS; Massimo Antonelli, MD, Study Chair — Fondazione Policlinico A. Gemelli IRCCS
Locations (11):
- Shamir Medical Center, Tel Aviv, Israel
- Italy (10):
  - Azienda ospedaliera universitaria "Ospedali riuniti di Ancona", Ancona
  - Azienda ospedaliera universitaria "Policlinico di Bari", Bari
  - Humanitas Research Hospital, Milan
  - Azienda ospedaliera universitaria di Modena, Modena
  - Azienda ospedaliera Federico II, Napoli
  - Azienda ospedaliera universitaria "Luigi Vanvitelli", Napoli
  - Policlinico "P. Giaccone", Palermo
  - Azienda ospedaliera Perugia, Perugia
  - Fondazione Policlinico "A. GEMELLI", Roma
  - Azienda ospedaliera universitaria Città della Salute e della Scienza di Torino - presidio Molinette, Torino